CLINICAL TRIAL: NCT03792633
Title: Phase 2 Study of Humanized CD19-directed Chimeric Antigen Receptor-modified T Cells (huCART19) for Very High-Risk Subsets of B Cell Acute Lymphoblastic Leukemia (B-ALL)
Brief Title: Study of huCART19 for Very High-Risk (VHR) Subsets of Pediatric B-ALL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Children's Hospital of Philadelphia (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 831916; 18CT014 (Other: CHOP)
Record Dates: First submitted 2019-01-02; First posted 2019-01-03 (Actual); Results first posted 2025-05-16 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-05

CONDITIONS: Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Newly Diagnosed VHR B-ALL or High-Risk Relapse of B (Experimental)
  Interventions: Biological: huCART19
- Poor Response to Prior B Cell Directed Engineered cell therapy (Experimental)
  Interventions: Biological: huCART19

INTERVENTIONS:
Biological: huCART19 — IV injection

SUMMARY:
This is a phase 2 study to evaluate humanized CD19 redirected autologous T cells (or huCART19 cells) with CD19 expressing relapsed and refractory B-cell acute lymphoblastic leukemia. This study is targeting pediatric and young adult patients aged 3 months - 29 years with CD19+ B cell malignancies in newly diagnosed B-ALL patients predicted to have an exceedingly poor outcome with conventional chemotherapy, in high-risk first relapse, or and in second or greater relapse in this phase 2 trial. In addition, a second cohort will test the efficacy of huCART19 in patients with poor response to prior B cell directed engineered cell therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent form must be obtained.
2. Relapsed or refractory B-cell ALL:

   a. Cohort A: Patients with newly diagnosed VHR B-ALL or high-risk relapse of B-ALL who meet one of the following criteria:

   i. Newly diagnosed NCI HR B-ALL with induction failure: M3 marrow (>25% blasts) at end of induction OR

ii. First marrow relapse of B-ALL at < 36 months from diagnosis OR iii. 2nd or greater relapse OR

iv. Any relapse after allogeneic HSCT and ≥ 4 months from SCT at enrollment OR

v. Refractory disease defined as having not achieved an MRD-negative and/or CSF-negative CR after ≥ 2 chemotherapy regimens/cycles of frontline therapy or 1 cycle of reinduction therapy for patients in first relapse OR

vi. Ineligible for allogeneic SCT because of:

1. Comorbid disease
2. Other contraindications to allogeneic SCT conditioning regimen
3. Lack of suitable donor
4. Prior SCT
5. Declines allogeneic SCT as the therapeutic option after documented discussion, with expected outcomes, about the role of SCT with a BMT physician not part of the study team b. Cohort B: Patients previously treated with B cell directed engineered cell therapy who meet one of the following criteria: i. partial response or no response to prior cell therapy ii. CD19+ relapse after prior cell therapy iii. demonstrated early (≤6 months from infusion) B cell recovery suggesting loss of engineered cells c. Patients with prior or current history of CNS3 disease will be eligible if CNS disease is responsive to therapy (at infusion, must meet criteria in Section 5.3 of the protocol)

3. Documentation of CD19 tumor expression in bone marrow, peripheral blood, CSF, or tumor tissue by flow cytometry at relapse (or a recent sample in the case of refractory disease). If the patient has received CD19-directed therapy, then the flow cytometry should be obtained after this therapy to show CD19 expression.

4. Adequate organ function defined as:

1. A serum creatinine based on age/gender
2. ALT≤ 500 U/L
3. Bilirubin ≤2.0 mg/dl
4. Must have a minimum level of pulmonary reserve defined as ≤ Grade 1 dyspnea, < Grade 3 hypoxia; DLCO ≥ 40% (corrected for anemia) if PFTs are clinically appropriate as determined by the treating investigator
5. Left Ventricular Shortening Fraction (LVSF) ≥ 28% or Ejection Fraction (LVEF) ≥ 45% confirmed by ECHO, or adequate ventricular function documented by a scan or a cardiologist.

   5. Age 3 months to 29 years. 6. Adequate performance status (Lansky or Karnofsky score ≥50). 7. Subjects of reproductive potential must agree to use acceptable birth control methods.

   Exclusion Criteria:
   1. Active hepatitis B or active hepatitis C.
   2. HIV Infection.
   3. Active acute or chronic graft-versus-host disease (GVHD) requiring systemic therapy.
   4. Concurrent use of systemic steroids or immunosuppression at the time of cell infusion or cell collection, or a condition, in the treating physician's opinion, that is likely to require steroid therapy or immunosuppression during collection or after infusion. Steroids for disease treatment at times other than cell collection or at the time of infusion are permitted. Use of physiologic replacement hydrocortisone or inhaled steroids is permitted as well.
   5. CNS3 disease that is progressive on therapy, or with CNS parenchymal lesions that might increase the risk of CNS toxicity.
   6. Pregnant or nursing (lactating) women.
   7. Uncontrolled active infection.
   8. Active medical disorder that, in the opinion of the investigator, would substantially increase the risk of uncontrollable CRS or neurotoxicity.

Ages: 3 Months to 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 106 (Actual)
Dates: Start 2019-01-18 (Actual); Primary Completion 2024-04-04 (Actual); Study Completion 2024-04-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shannon Maude, MD, PhD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Pennsylvania, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort A: Newly Diagnosed VHR B-ALL or High-Risk Relapse of B
- Cohort B: Poor Response to Prior B Cell Directed Engineered cell therapy
Period: Overall Study
Arm/Group | Cohort A | Cohort B
Started | 55 | 51
Completed | 26 | 21
Not Completed | 29 | 30
Not completed — Alternative Treatment | 17 | 19
Not completed — Death | 2 | 0
Not completed — Disease progression | 8 | 9
Not completed — Lost to Follow-up | 1 | 1
Not completed — Screen fail | 1 | 0
Not completed — Second malignancy | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A | Cohort B | Total
Number analyzed (Participants) | 55 | 51 | 106
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 43 | 44 | 87
  Between 18 and 65 years | 12 | 7 | 19
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 12.0 [1 to 29] | 11.6 [0.9 to 28] | 11.8 [0.9 to 29]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 25 | 45
  Male | 35 | 26 | 61
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 2 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 2 | 5
  White | 28 | 40 | 68
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 21 | 7 | 28

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Event-Free Survival in Patients With Newly Diagnosed VHR B-ALL or High-risk Relapse of B-ALL 1 Year After Treatment.
Description: Time from infusion to the first of event or censoring Events = Relapse, No Response, or Death; Censoring =Initiation of New Anticancer Therapy, Last Day of Follow-up/EOS; whichever occurs first.
Time Frame: 1 year
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Groups:
- Cohort A: Patients with newly diagnosed VHR B-ALL or high-risk relapse of B-ALL
Arm/Group | Cohort A
Number analyzed (Participants) | 52
percentage of subjects | 68.9 [56.8 to 83.5]

2. Primary Outcome: Number of Subjects With Event-Free Survival in Patients With Poor Response to Prior B Cell Directed Engineered Cell Therapy 1 Year After Treatment.
Description: Time from infusion to the first of event or censoring Events = Relapse, No Response (including CR/CRi without B Cell Aplasia), or Death; Censoring =Initiation of New Anticancer Therapy, Last Day of Follow-up/EOS; whichever occurs first.
Time Frame: 1 year
Measure: Number (95% Confidence Interval); unit: percentage of subject
Arm/Group | Cohort B
Number analyzed (Participants) | 48
percentage of subject | 62 [49 to 78.4]

3. Secondary Outcome: Overall Remission Rate
Description: Overall remission rate as determined by the response at day 28, computed as the number of subjects with CR or Cri, in patients with newly diagnosed VHR B-ALL or high-risk relapse of B-ALL.
Time Frame: 28 Days
Measure: Count of Participants; unit: Participants
Groups:
- Cohort B: Patients with poor response to prior B cell directed engineered cell therapy
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 52 | 48
Participants | 46 | 43

4. Secondary Outcome: Overall Remission Rate (Cohort B)
Description: Number of subjects with CR/CRi with B Cell Aplasia at Day 28
Time Frame: 28 Days
Population: Only subjects in cohort B analyzed in this measurement
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort B
Number analyzed (Participants) | 48
Participants | 37

5. Secondary Outcome: Percentage of Subjects With Relapse-free Survival
Description: Time from first response of CR/CRi to the first of event or censoring, in responders.
  Cohort A: Events = Relapse or Death; Censoring = Initiation of New Anticancer Therapy, Last Day of Follow-up/EOS; whichever occurs first.
  Cohort B: When defining responders, CR/CRi without B Cell Aplasia is considered no response. Events = Relapse or Death; Censoring = Initiation of New Anticancer Therapy, Last Day of Follow-up/EOS; whichever occurs first.
Time Frame: 1 year
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 52 | 48
percentage of subjects | 76.3 [64.3 to 90.4] | 80.4 [67.4 to 95.4]

ADVERSE EVENTS:
Time Frame: 1 year
Description: Adverse events were collected from only those subjects who were given the intervention.
Arm/Group | Cohort A | Cohort B
All-Cause Mortality (participants affected / at risk) | 2/55 | 0/51
Serious Adverse Events (participants affected / at risk) | 45/52 | 32/48
Other Adverse Events (participants affected / at risk) | 52/52 | 46/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A (N=52) | Cohort B (N=48)
Febrile neutropenia (Blood and lymphatic system disorders) | 37 (65) | 27 (35)
Left ventricular systolic dysfunction (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Eye disorders - Other (Right soft tissue orbital mass) (Eye disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Esophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal disorders - Other (Gastrointestinal hemorrhage) (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
Chills (General disorders) | 1 (1) | 0 (0)
Fever (General disorders) | 15 (18) | 9 (10)
Pain (General disorders) | 1 (1) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cytokine release syndrome (Immune system disorders) | 44 (62) | 28 (35)
Catheter related infection (Infections and infestations) | 2 (2) | 1 (1)
Infections and infestations - Other (Bacterial infectious disorder) (Infections and infestations) | 1 (2) | 0 (0)
Infections and infestations - Other (Disseminated fungal infection) (Infections and infestations) | 1 (1) | 0 (0)
Infections and infestations - Other (Metapneumovirus) (Infections and infestations) | 1 (1) | 0 (0)
Infections and infestations - Other (RSV) (Infections and infestations) | 1 (1) | 0 (0)
Infections and infestations - Other (S. epidermidis) (Infections and infestations) | 1 (1) | 0 (0)
Infections and infestations - Other (SARS-CoV-2) (Infections and infestations) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 3 (3) | 0 (0)
Myelitis (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 4 (4) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 1 (1)
Vascular access complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 3 (3) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1)
Creatinine increased (Investigations) | 3 (3) | 1 (1)
Electrocardiogram QT corrected interval prolonged (Investigations) | 0 (0) | 1 (1)
Fibrinogen decreased (Investigations) | 5 (6) | 1 (1)
INR increased (Investigations) | 5 (5) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Bone Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Dysphasia (Nervous system disorders) | 1 (1) | 0 (0)
Edema cerebral (Nervous system disorders) | 1 (1) | 1 (1)
Encephalopathy (Nervous system disorders) | 4 (4) | 0 (0)
Headache (Nervous system disorders) | 3 (4) | 2 (2)
Nervous system disorders - Other (CAR Neurotoxicity) (Pregnancy, puerperium and perinatal conditions) | 13 (14) | 7 (7)
Seizure (Nervous system disorders) | 1 (1) | 2 (3)
Tremor (Nervous system disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Laryngeal edema (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Laryngeal stenosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (2)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 10 (10) | 3 (3)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 10 (10) | 2 (3)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A (N=52) | Cohort B (N=48)
Sinus bradycardia (Cardiac disorders) | 3 (5) | 3 (5)
Ear Pain (Ear and labyrinth disorders) | 3 (4) | 1 (1)
Blurred vision (Eye disorders) | 2 (3) | 3 (5)
Photophobia (Eye disorders) | 3 (3) | 1 (2)
Anemia (Blood and lymphatic system disorders) | 43 (119) | 37 (79)
Sinus tachycardia (Cardiac disorders) | 26 (60) | 24 (50)
Abdominal pain (Gastrointestinal disorders) | 16 (28) | 11 (14)
Constipation (Gastrointestinal disorders) | 9 (12) | 13 (20)
Diarrhea (Gastrointestinal disorders) | 15 (29) | 10 (22)
Nausea (Gastrointestinal disorders) | 38 (105) | 24 (48)
Oral hemorrhage (Gastrointestinal disorders) | 2 (4) | 3 (3)
Oral pain (Gastrointestinal disorders) | 5 (5) | 2 (2)
Vomiting (Gastrointestinal disorders) | 37 (115) | 22 (60)
Chills (General disorders) | 8 (10) | 2 (4)
Fatigue (General disorders) | 38 (76) | 34 (54)
Fever (General disorders) | 14 (19) | 12 (17)
Generalized edema (General disorders) | 3 (6) | 2 (4)
Pain (General disorders) | 21 (39) | 18 (29)
Cytokine release syndrome (Immune system disorders) | 6 (6) | 11 (11)
Immune system disorders - Other (Hypogammaglobulinemia) (Immune system disorders) | 28 (75) | 25 (55)
Infections and infestations - Other (Influenza) (Infections and infestations) | 0 (0) | 3 (3)
Infections and infestations - Other (Rhinovirus) (Infections and infestations) | 0 (0) | 3 (6)
Infections and infestations - Other (SARS-CoV-2) (Infections and infestations) | 5 (7) | 12 (17)
Papulopustular rash (Infections and infestations) | 3 (3) | 2 (2)
Sinusitis (Infections and infestations) | 6 (15) | 5 (15)
Skin infection (Infections and infestations) | 0 (0) | 3 (7)
Upper respiratory infection (Infections and infestations) | 8 (16) | 4 (7)
Bruising (Injury, poisoning and procedural complications) | 11 (14) | 13 (17)
Injury, poisoning and procedural complications - Other (Bone marrow aspiration site pain) (Injury, poisoning and procedural complications) | 4 (10) | 7 (9)
Injury, poisoning and procedural complications - Other (Bug bite) (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Vascular access complication (Injury, poisoning and procedural complications) | 4 (7) | 1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 28 (84) | 33 (88)
Alanine aminotransferase increased (Investigations) | 13 (37) | 17 (42)
Aspartate aminotransferase increased (Investigations) | 15 (36) | 12 (39)
Blood bilirubin increased (Investigations) | 8 (16) | 3 (7)
Creatinine increased (Investigations) | 13 (30) | 7 (15)
INR increased (Investigations) | 20 (52) | 15 (24)
Lymphocyte count decreased (Investigations) | 44 (174) | 43 (152)
Neutrophil count decreased (Investigations) | 46 (249) | 40 (208)
Platelet count decreased (Investigations) | 37 (119) | 31 (73)
White blood cell decreased (Investigations) | 47 (187) | 43 (165)
Anorexia (Metabolism and nutrition disorders) | 41 (102) | 27 (55)
Dehydration (Metabolism and nutrition disorders) | 4 (6) | 2 (4)
Hyperglycemia (Metabolism and nutrition disorders) | 9 (21) | 3 (9)
Hyperphosphatemia (Metabolism and nutrition disorders) | 2 (6) | 15 (22)
Hyperuricemia (Metabolism and nutrition disorders) | 11 (17) | 8 (8)
Hypocalcemia (Metabolism and nutrition disorders) | 5 (11) | 2 (9)
Hypokalemia (Metabolism and nutrition disorders) | 11 (36) | 6 (21)
Hyponatremia (Metabolism and nutrition disorders) | 2 (5) | 3 (9)
Hypophosphatemia (Metabolism and nutrition disorders) | 2 (6) | 5 (9)
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 (8) | 3 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 7 (11) | 6 (17)
Bone pain (Musculoskeletal and connective tissue disorders) | 4 (5) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 3 (4) | 2 (3)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 3 (6) | 2 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 19 (32) | 15 (24)
Neck pain (Musculoskeletal and connective tissue disorders) | 4 (5) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 15 (30) | 10 (13)
Dizziness (Nervous system disorders) | 13 (16) | 6 (9)
Headache (Nervous system disorders) | 37 (105) | 31 (63)
Lethargy (Nervous system disorders) | 3 (3) | 1 (1)
Tremor (Nervous system disorders) | 8 (11) | 6 (6)
Agitation (Psychiatric disorders) | 7 (11) | 0 (0)
Anxiety (Psychiatric disorders) | 4 (7) | 3 (4)
Confusion (Psychiatric disorders) | 8 (10) | 5 (5)
Hallucinations (Psychiatric disorders) | 4 (5) | 1 (1)
Insomnia (Psychiatric disorders) | 7 (8) | 4 (8)
Irritability (Psychiatric disorders) | 4 (4) | 3 (4)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 3 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 27 (45) | 16 (19)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 9 (24) | 6 (10)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 4 (11) | 2 (4)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 10 (14) | 9 (13)
Respiratory, thoracic and mediastinal disorders - Other (Tachypnea) (Respiratory, thoracic and mediastinal disorders) | 3 (7) | 5 (10)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 16 (20) | 7 (8)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 7 (8) | 5 (6)
Eczema (Skin and subcutaneous tissue disorders) | 6 (8) | 3 (5)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (2) | 3 (4)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 4 (5)
Pruritus (Skin and subcutaneous tissue disorders) | 9 (11) | 6 (10)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 18 (32) | 13 (16)
Skin and subcutaneous tissue disorders - Other (Rash) (Skin and subcutaneous tissue disorders) | 3 (6) | 3 (4)
Hot flashes (Vascular disorders) | 3 (4) | 0 (0)
Hypertension (Vascular disorders) | 4 (7) | 1 (3)
Hypotension (Vascular disorders) | 12 (28) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-08-19): https://cdn.clinicaltrials.gov/large-docs/33/NCT03792633/Prot_SAP_000.pdf
  • Informed Consent Form (2023-08-11): https://cdn.clinicaltrials.gov/large-docs/33/NCT03792633/ICF_001.pdf